CLINICAL TRIAL: NCT02587247
Title: Apport de l'Immuno-TEP préciblée Avec l'Anticorps bispécifique Anti-ACE x Anti-HSG TF2 et le Peptide IMP-288 marqué au Gallium-68 Pour l'Imagerie Des Patients Potentiellement Candidats à Une Chirurgie d'exérèse et/ou Thermoablation Locale d'Une ou Plusieurs métastases, au Diagnostic ou Lors de la Rechute de Cancers Colo-rectaux (CCR) Exprimant l'antigène Carcino-embryonnaire (ACE): Comparaison au Bilan Conventionnel
Brief Title: ImmunoTEP With 68-Ga in Metastatic Colo Rectal Cancer
Acronym: iTEP Colon
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC14_0428
Record Dates: First submitted 2015-10-19; First posted 2015-10-27 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TF2 antibody/68Ga-IMP-288 (Experimental): TF2 antibody/68Ga-IMP-288
  Interventions: Drug: TF2 antibody/68Ga-IMP-288

INTERVENTIONS:
Drug: TF2 antibody/68Ga-IMP-288 — TF2 antibody coupled with 68Ga-IMP-288

SUMMARY:
Evaluation of the sensitivity of the immuno-PET PET / CT pretargeted with the bispecific anti-CEA x anti-HSG TF2 antibody and IMP-288 peptide labeled with Gallium-68 for imaging potential candidate patients for surgery of local resection of one or more metastases at diagnosis or during relapse CCR expressing CEA.

DETAILED DESCRIPTION:
Injection of a bispecific anti-CEA x anti-HSG antibody TF2 (120 nmoles) and 30 hours later IMP-288 peptide labeled with gallium-68 (3 to 6 nmoles/150 MBq). A TEP imaging acquisition is plannified 60 min after the 68-Ga injection.

ELIGIBILITY:
Inclusion Criteria:

* Existence of one or more metastases of of colorectal cancer (CRC) expressing the CEA , potentially accessible by surgical or thermo resection at the moment of the diagnosis or at relapse.

OR

* Isolated and progressive elevation of plasma CEA during the monitoring of CRC with high metastatic risk
* More than 18 years
* Negative pregnancy test for women of childbearing age. Women of childbearing age should take effective continuous contraception for 3 months.
* At least 4 weeks after the last treatment and after recovery of potential toxicity
* Karnofsky more than 70 or ECOG 0-1
* Life expectancy of at least 6 months
* CEA positive immunohistochemistry or plasma CEA supperior or equal to the normal level
* Creatinin less or equal 200 micromol/L
* Signed informed consent
* geographical proximity

Exclusion Criteria:

* Pregnancy or breastfeeding
* Serious illness or comorbidity assessed risk
* History of other cancer within 5 years, with the exception of skin carcinomas other than melanomas or in-situ carcinoma of the cervix
* Anti-antibody presence in patients who have already received antibody
* Hypersensitivity to antibodies or proteins
* Intellectual inability to sign the informed consent
* Insulin-dependent diabetic patient or non-insulin dependent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the sensitivity of the immuno-PET PET / CT pretargeted with the bispecific anti-CEA x anti-HSG TF2 antibody and IMP-288 peptide labeled with Gallium-68 | Month 3
  Initial and M3 imaging assessment comparaison, and/or immunohistochemistry

SECONDARY OUTCOMES:
To compare the diagnostic performance of immuno-PET with morphological and functional imaging procedures currently performed in the imaging assessment (CT, ultrasound + liver MRI, FDG-PET). | Month 3
  Identified lesions at initial and M3 imaging assessment will be compared with lesions identified with 68-Ga-PET
To Determine the value of immuno-PET in terms of specificity and predictive value. This determination will be made at the "patient" and at the "injury level. | Month 3
  Comparaison with baseline imaging assessment, Month 3 imaging and/or immunohistochemistry evaluation
To assess the safety of the procedure | Month 3
  Biological and clinical examen of the patients between Day 1 and month 3 follow up. The assement will be according to NCI criteria
Search for the development of a blood Immunization against the products | Month 3
  Human anti Human antibody test by immuno assay at base line, M1 and M3
To study the expression of CEA intensity on surgical excision parts in surgical patients and compare it to the semi-quantitative immuno-PET | No more than 3 months (it depend of the day of the surgery)
  Immunohistochemistry analysis with anti CEA antibody
To evaluate the clinical impact (new lecture of imaging, new examens) | M1
  A form will be fill in by the physican who request the immuno PET

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU, Nantes
  - Institut de cancérologie de l'Ouest, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Touchefeu Y, Bailly C, Frampas E, Eugene T, Rousseau C, Bourgeois M, Bossard C, Faivre-Chauvet A, Rauscher A, Masson D, David A, Cerato E, Carlier T, Sharkey RM, Goldenberg DM, Barbet J, Kraeber-Bodere F, Bodet-Milin C. Promising clinical performance of pretargeted immuno-PET with anti-CEA bispecific antibody and gallium-68-labelled IMP-288 peptide for imaging colorectal cancer metastases: a pilot study. Eur J Nucl Med Mol Imaging. 2021 Mar;48(3):874-882. doi: 10.1007/s00259-020-04989-3. Epub 2020 Aug 21. PMID 32820369